CLINICAL TRIAL: NCT01191996
Title: A Phase 2, Open-label, Dose-escalation Study Evaluating the Safety, Tolerability, and Pharmacodynamics of Intravenously Administered MIS416 in Patients With Chronic Progressive Multiple Sclerosis
Brief Title: Safety Study of an Immunomodulating Microparticle to Treat Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innate Immunotherapeutics (Industry)
Collaborators: Primorus Clinical Trials (Unknown); National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIS416-201
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis
Keywords: SPMS; PPMS; MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — MIS416 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIS416 (Experimental): MIS416, immunomodulating microparticle, given intravenously weekly
  Interventions: Biological: MIS416

INTERVENTIONS:
Biological: MIS416 — MIS416 intravenously every week

SUMMARY:
The purpose of the study is to determine the safety and tolerability, dose-limiting toxicities, maximum tolerated dose, and recommended therapeutic dose of intravenously administered MIS416 weekly in patients with chronic progressive multiple sclerosis.

DETAILED DESCRIPTION:
This is a single center, open-label, non-randomized, dose-escalation study, to be conducted in two phases:

* a dose-escalation (DE) phase, to evaluate the safety, tolerability, MTD, and PD of MIS416 administered IV once weekly for 4 doses; and
* a dose-confirmation (DC) phase, which will be a cohort expansion at or below the MTD (i.e., the RTD) of MIS416, dosed once weekly for up to 12 doses.

Subjects will be treated with a weekly IV dose of MIS416 in 28-day cycles: 1 cycle in the DE phase, and up to 3 cycles in the DC phase. Subjects will be evaluated and dosed weekly each cycle in each phase. Subjects will return for a follow-up visit 7 days after completion of the last dose of study drug.

The primary objectives of this study are:

1. To determine the safety and tolerability, dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended therapeutic dose (RTD) of intravenously (IV) administered MIS416 weekly in patients with chronic progressive multiple sclerosis (CPMS); and
2. To assess the pharmacodynamic (PD) effects of MIS416, including effects on serum cytokine levels and peripheral blood mononuclear cell (PBMC) composition, cytokine/chemokine expression and function.

The secondary objectives of this study are:

1. To document any changes in MS clinical status occurring during the 12-week MIS416 dosing period in the dose-confirmation phase, as determined by the Multiple Sclerosis Functional Composite (MSFC), Fatigue Severity Scale (FSS), Short Form Health Survey (SF-36), and Expanded Disability Status Scale (EDSS); the frequency of clinical relapses; and signs of clinical activity on serial cranial MRI scans; and
2. To evaluate, in exploratory fashion, any correlations between clinical, radiological and PD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Diagnosis of MS, by the McDonald criteria.
* Chronic progressive MS (CPMS), defined as either primary progressive MS (PPMS) or secondary progressive MS (SPMS), per the criteria of the National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. [NOTE: In the dose-confirmation phase, only subjects with SPMS may be enrolled].
* MS is clinically active with worsening clinical status within the past 2 years, defined as an increase in EDSS by 1 point or more, sustained for at least 6 months.
* Expanded Disability Status Scale (EDSS) of 2.5 to 7.0 at Screening.
* The following laboratory values must be documented within 3 days prior to initiation of study drug:

  * Absolute neutrophil count (ANC) >= 1 x 109/L
  * Platelet count >= 100 x 109/L
  * Serum creatinine =< 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) =< 2 × upper limit of normal.
* Provide written informed consent to participate.

Exclusion Criteria:

* Relapsing-remitting MS or progressive-relapsing MS
* Any immunomodulatory drug therapy or immunosuppressive therapy within the previous six months, or vaccine or systemic corticosteroids within the previous 60 days, prior to initiation of study drug.
* Exposure to other experimental treatments currently under investigation in MS clinical trials, including alemtuzamab, rituximab, fingolimod, and clabribine.
* A diagnosis or history of collagen vascular disease (including Sjögren's syndrome and systemic lupus erythematosus), anticardiolipin antibody syndrome, cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL), sarcoidosis, vasculitis, Bechet's syndrome and/or Lyme disease.
* History of alcohol or drug abuse (with the exception of cannabinoids) within 2 years prior to initiation of study drug.
* Previous exposure to MIS416.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety profile, including maximum tolerated dose | 1 month in DE phase, 3 months in DC phase
  Dose-limiting toxicities, adverse events, safety MRI assessments

SECONDARY OUTCOMES:
Pharmacodynamic assessments | 1 month in DE phase, 3 months in DC phase
  Serum and cellular immunological assays
MRI assessments | 1 month in DE phase, 3 months in DC phase
  Safety MRIs
Clinical status | 3 months in DC phase
  Neurological examination, Expanded Disability Status Scale (EDSS), Multiple Sclerosis Functional Composite (MSFC), Fatigue Severity Scale (FSS), Multiple Sclerosis Quality of Life (MSQLI).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Luckey, Principal Investigator — Primorus Clinical Trials; Tim Anderson, Principal Investigator — Department of Medicine, University of Otago
Locations (1):
- Primorus Clinical Trials, 40 Stewart Street, Christchurch, Canterbury, New Zealand

REFERENCES:
- [Derived] Webster GA, Sim DA, La Flamme AC, Mayo NE. Evaluation of neurological changes in secondary progressive multiple sclerosis patients treated with immune modulator MIS416: results from a feasibility study. Pilot Feasibility Stud. 2017 Nov 16;3:60. doi: 10.1186/s40814-017-0201-4. eCollection 2017. PMID 29177070
- [Derived] Luckey AM, Anderson T, Silverman MH, Webster G. Safety, tolerability and pharmacodynamics of a novel immunomodulator, MIS416, in patients with chronic progressive multiple sclerosis. Mult Scler J Exp Transl Clin. 2015 May 12;1:2055217315583385. doi: 10.1177/2055217315583385. eCollection 2015 Jan-Dec. PMID 28607691